CLINICAL TRIAL: NCT03065413
Title: The PrOspeCtive HEllenic NAval PersoNnel StUdy in CardiovaScular Diseases (OCEANUS Study)
Brief Title: It is a Prospective Study Aiming to Identify Incidence and Prevalence of Cardiovascular Diseases, Changes in Physical Activity, Dietary Habits and Anxiety Depression Levels Through a Period of Time in the Naval Personnel (PrOspeCtive HEllenic NAval PersoNnel StUdy in CardiovaScular Diseases)
Acronym: OCEANUS
Status: Recruiting | Type: Observational
Sponsor: Naval Hospital, Athens (Other)
Responsible Party: Principal Investigator, MASTROKOSTOPOULOS ANTONIOS, Consultant Cardiologist, Naval Hospital, Athens
Other Study IDs: F.700/28/165531/S.2743
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Cardiovascular Diseases; Risk Factor, Cardiovascular
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective study. Starting from 2014 all newly appointed 1st year cadets in Naval Academies will be enrolled until the class of 2025.

Physical examination, food frequency questionnaire, physical activity questionnaire, anxiety/depression questionnaire, medical history will be filled out at first interview.

Specific blood tests will be performed. Every participant will be interviewed every three years and will complete the same questionnaires.

Follow up period is determined ten years after last class enrollment

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Non signed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Incidence / prevalence of CVD | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Aikaterini Roumpi, MD MSc, Principal Investigator — Athens Naval Hospital
Locations (1):
- Athens Naval Hospital, Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided